CLINICAL TRIAL: NCT02899364
Title: Groningen Intervention Study for the Preservation of Cardiac Function With Sodium Thiosulfate After ST-segment Elevation Myocardial Infarction
Brief Title: Sodium Thiosulfate to Preserve Cardiac Function in STEMI
Acronym: GIPS-IV
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Pim van der Harst, MD, PhD, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: GIPS-IV; 2015-001006-34 (EudraCT Number)
Record Dates: First submitted 2016-08-31; First posted 2016-09-14 (Estimated); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Myocardial Infarction; Heart Failure
Keywords: Sodium thiosulfate; STEMI; Infarct size; Cardiac magnetic resonance imaging; Hydrogen sulfide
MeSH Terms: conditions — Myocardial Infarction; Heart Failure; ST Elevation Myocardial Infarction | interventions — sodium thiosulfate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium thiosulfate (Experimental): 25 gram sodium thiosulfate is given intravenously in two doses of 12.5 gram (50mL) dissolved in 250 ml sodium chloride 0.9%. Upon arrival at the cath-lab, after confirming in- and exclusion criteria and obtaining verbal informed consent the first dose, will be administered in 20 minutes (infusion rate 15 mL/min). After infusion the patient will receive primary percutaneous coronary intervention. Post-PCI the patient will be admitted to the coronary care unit where he will receive the second dose, 6 hours after start of the first dose. The second dose is administered in 30 minutes (infusion rate 10 mL/min). At 4 months infarct size is assessed by LGE cardiac magnetic resonance imaging.
  Interventions: Drug: Sodium thiosulfate; Procedure: primary percutaneous coronary intervention; Other: cardiac magnetic resonance imaging
- Sodium chloride 0.9% (Placebo Comparator): 50 ml Sodium chloride 0.9%, added to 250ml sodium chloride 0.9% is administered twice. Upon arrival at the cath-lab, after confirming in- and exclusion criteria and obtaining verbal informed consent the first dose, will be administered in 20 minutes (infusion rate 15ml/min). After infusion the patient will receive primary percutaneous coronary intervention. Post-PCI the patient will be admitted to the coronary care unit where he receive the second dose, 6 hours after start of the first dose. The second dose is administered in 30 minutes (infusion rate 10 mL/min). At 4 months infarct size is assessed by LGE cardiac magnetic resonance imaging.
  Interventions: Drug: Sodium chloride 0.9%; Procedure: primary percutaneous coronary intervention; Other: cardiac magnetic resonance imaging

INTERVENTIONS:
Drug: Sodium thiosulfate — see description under experimental arm
  Arms: Sodium thiosulfate
Drug: Sodium chloride 0.9% — see description under placebo comparator arm
  Other Names: Placebo
  Arms: Sodium chloride 0.9%
Procedure: primary percutaneous coronary intervention — Primary treatment of the ischemia-related coronary artery is left to discretion of the operator and might consist of thrombus aspiration, balloon inflation and stent implantation. Additional balloon angioplasty or stenting of the culprit or other lesions will be performed when necessary.
  Other Names: PPCI
Other: cardiac magnetic resonance imaging — CMR-imaging will be used for assessment of infarct size, left ventricular function, quantification of myocardial scar and diffuse myocardial fibrosis. CMR-imaging examinations will be performed on a 3 Tesla scanner using a phased array cardiac receiver coil at 4 months after randomization according to standard protocols. The full study protocol lasts approximately 45 minutes and includes anatomy and function, LGE and T1-mapping.
  Other Names: CMR-imaging

SUMMARY:
Rationale: Timely and effective reperfusion by primary percutaneous coronary intervention (PPCI) is currently the most effective treatment of ST-segment elevation myocardial infarction (STEMI). However, permanent myocardial injury related to the ischemia and subsequent reperfusion is observed in the vast majority (88%) of patients and harbours a risk of heart failure development. Administration of hydrogen sulfide (H2S) has been shown to protect the heart from "ischemia reperfusion injury" in various experimental models. Data in humans suggests that the H2S-releasing agent sodium thiosulfate (STS) can be administered safely.

Objective: to evaluate the efficacy and safety of STS compared to placebo treatment on myocardial infarct size in patients presenting with STEMI and treated with PCI

Study design: a multicenter, double blind, randomized controlled clinical trial. A total of 380 patients, aged 18 years and above, undergoing primary PCI for a first STEMI and deemed amenable, by the investigator, to be treated with STS 12.5g intravenously (i.v.) or matched placebo immediately after arrival at the catheterization laboratory (cath-lab) and a repeated dose administered 6 hours after the first dose, on top of standard treatment. Primary endpoint is infarct size as measured with cardiac magnetic resonance imaging (CMR-imaging) 4 months after randomization.

DETAILED DESCRIPTION:
Introduction and rationale:

Despite the recent advances in treatment, acute myocardial infarction (AMI) frequently results in permanent myocardial injury imposing an increased risk for adverse cardiac remodelling, diminished cardiac function and the development of heart failure. Decreased cardiac function after PPCI is associated with impaired prognosis. In addition to PPCI, cornerstones pharmacological treatment of myocardial infarction (MI) includes; (1) treatment direct against blood coagulation with platelet aggregation inhibitors, (2) cholesterol lowering treatment with statins; (3) sympathicus inhibition by beta-blocker treatment; and (4) inhibitors of the renin-angiotensin-aldosterone system. These therapies were successfully implemented over the last decades and resulted in substantial improvements of prognosis after AMI.

Although timely PPCI has a tremendous benefit in AMI, not only ischemia but also reperfusion itself is considered to cause myocardial injury and cardiomyocyte death. This phenomena is referred to as "ischemia reperfusion injury" in literature and is caused by the sudden restoration of blood flow and its accompanying intracellular acidity (pH) change and calcium overload, cardiomyocyte hypercontracture, myocardial inflammation, oxidative stress generation and mitochondrial permeability transition pore opening. Reducing ischemia reperfusion injury is expected to further decrease infarct size, decreasing adverse cardiac remodelling and improving cardiac function as well as clinical outcome.

The investigators expect a substantial beneficial effect of H2S in the prevention of ischemia reperfusion injury. H2S is the third endogenous gaseous transmitter next to carbon monoxide (CO) and nitric oxide (NO) and is involved as a physiological mediator in several body organ and tissue processes. H2S is synthesized endogenously by enzymatic and non-enzymatic pathways. A non-enzymatic pathway is by the reductive reaction with thiosulfate, with pyruvate acting as a hydrogen donor. Thiosulfate itself acts as an intermediate in the sulfur metabolism of cysteine and is known as a metabolite of H2S and in that way also able to produce H2S, especially under hypoxic conditions.

H2S has been shown to protect from myocardial ischemia reperfusion injury in various experimental animal models; e.g. it reduces infarct size and apoptosis and attenuates cardiac function. Inhibition of leukocyte endothelial cell interactions, neutralization of reactive oxygen species (ROS) and the reduction of apoptotic signalling are the suggested as additional mechanisms underlying the cardioprotective effect of H2S. H2S has been shown to attenuate myocardial ischemia reperfusion in cellular, rodents and porcine animal models. H2S can be safely administered intravenously as STS to humans. STS has been demonstrated to detoxify cyanide poisoning in 1895 in dogs, is used in humans since 1933 for the treatment of cyanide intoxication, is used since the eighties for treatment of vascular calcifications in end-stage renal disease, and is used to prevent toxicity of cisplatin treatment. More recently, studies have shown STS can delay the progression of coronary artery calcification in haemodialysis patients. The aim of the GIPS-IV trial is to evaluate the efficacy and safety of STS compared to placebo treatment on myocardial infarct size in patients presenting with STEMI undergoing PPCI in a double blind randomized controlled clinical trial.

Study design:

The GIPS-IV trial is a multicenter, randomized, placebo-controlled, double blind trial. A total of 380 patients presenting with a first STEMI will be included. All patients will be randomly assigned, in a 1:1 ratio, to receive STS (12.5 mg iv) or matching placebo. Study medication will be administered twice. The first dose of study medication will be administered immediately after checking inclusion and exclusion criteria and obtaining verbal informed consent at the cath-lab. The second dose of study medication will be administered 6 hours later, at the Coronary Care Unit (CCU). The study will take place at the University Medical Centre of Groningen (UMCG), University Medical Center Utrecht (UMCU) and Treant Scheper hospital in Emmen, all high-volume centers with experience in care and research of patients with STEMI. The primary endpoint will be based on infarct size as measured by late gadolinium enhancement cardiac magnetic resonance imaging (LGE CMR)-imaging 4 months after STEMI, a period in which the remodelling of the heart is expected to be completed. LGE CMR-imaging is a well-recognized, validated, and highly reproducible technique. Total follow-up duration of the GIPS-IV trial is 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* The diagnosis STEMI defined by (1.) chest pain suggestive for myocardial ischemia for at least 30 minutes, the time from onset of the symptoms less than 12 hours before hospital admission, and (2.) an electrocardiogram (ECG) recording with ST- segment elevation of more than 0.1 millivolt (mV) in 2 or more contiguous leads or presence of new left bundle branch block;
* Symptoms and/or ST-segment deviation should be present (persisting) at time of arrival in the cath-lab;
* Primary PCI is being considered as treatment;
* Patient is willing to cooperate with follow-up during 2 years.

Exclusion Criteria:

* Prior MI (STEMI/non-STEMI/acute coronary syndrome (ACS), unless maximum troponin T < 50ng/L.
* Prior CABG;
* Prior PCI, complicated by periprocedural infarction, unless maximum troponin T < 50 ng/L;
* Known cardiomyopathy;
* Previous hospitalization for heart failure;
* Active malignancy (requiring chemotherapy, radiation or surgery at the time of randomization), except for adequately treated non-melanoma skin cancer or other noninvasive or in situ neoplasm (e.g., cervical cancer in situ);
* History of chemotherapy;
* History of radiotherapy in chest region;
* Relieve of symptoms and complete ST-segment resolution prior to arrival at the cath-lab;
* Known permanent atrial fibrillation;
* Presentation with cardiogenic shock (systolic blood pressure <90 mmHg);
* Severe hypertension (systolic blood pressure >220 mmHg);
* Sedated and/or intubated patients;
* The existence of a condition with a life expectancy of less than 1 year;
* Contraindication for 3 Tesla (T) CMR-imaging (e.g. body weight >150kg; known claustrophobia; 3 T magnetic resonance imaging (MRI) incompatible ferromagnetic objects in the body, end-stage renal disease);
* Pregnancy or breastfeeding women; women of childbearing potential with clinical suspicion of possible pregnancy;
* A condition which, according to the clinical judgment of the investigator and/or treating physician, does not allow the patient to successfully participate in the study.
* Contraindication for metoclopramide (e.g. Parkison; epilepsy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2018-07-20 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Myocardial infarct size as measured with late gadolinium enhancement cardiac magnetic resonance imaging. | 4 months after randomization
  Primary efficacy parameter

SECONDARY OUTCOMES:
Left ventricular ejection fraction as assessed by cardiac magnetic resonance imaging | 4 months after randomization
  Secondary efficacy parameter
N-terminal prohormone of brain natriuretic peptide (NT-proBNP) level (ng/L) | 4 months after randomization
  Secondary efficacy parameter
All cause mortality | 4 months after randomization and after 2-year follow-up
  Safety parameter
Combined major adverse cardiovascular events | 4 months after randomization and after 2-year follow-up
  Safety parameter. Includes cardiovascular mortality, re-infarction, re-intervention (any revascularization not planned on index CAG).
Incidence of stroke | 4 months after randomization and after 2-year follow-up
  Safety parameter. Cerebrovascular accident (both ischemic and non-ischemic).
Incidence of stent thrombosis | 4 months after randomization and after 2-year follow-up
  Safety parameter. Stent thrombosis confirmed with angiography.
Incidence of Implantable Cardioverter Defibrillator implantation | 4 months after randomization and after 2-year follow-up
  Safety parameter
Hospitalization for heart failure or chest pain | 4 months after randomization and after 2-year follow-up
  Safety parameter. defined as an overnight stay, with different dates for admission and discharge
Enzymatic infarct size as assessed by peak creatinine kinase myocardial band (CK-MB). | 0-3 days after randomization (during hospitalization)
  Safety parameter

OTHER OUTCOMES:
Health related quality of life: EuroQol EQ-5D-5L | 0-5 days after randomization (during hospitalization) and at 4 months follow up
  Health related quality of life assessed using the EuroQol EQ-5D-5L.
  The EQ-5D-5L has 2 components:
  There is a descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, unable/extreme problems. The respondent is asked to indicate his/her health state by ticking (or placing a cross) in the box against the most appropriate statement in each of the 5 dimensions.
  The EQ VAS records the respondent's self-rated health on a 20 cm vertical, visual analogue scale with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine'.
  The users guide gives details of the scoring system: https://euroqol.org/wp-content/uploads/2016/09/EQ-5D-5L_UserGuide_2015.pdf
General affective status | 0-5 days after randomization (during hospitalization) and at 4 months follow up
  Assessed with PANAS questionnaire (Positive And Negative Affect Schedule), positive affect score can range from 10 to 50, with higher scores representing higher positive affective state; negative affect score ranges from 10 to 50 with lower scores representing lower levels of negative affect
Creatine Kinase (U/L) | 0-3 days after randomization (during hospitalization)
  Changes in blood biomarkers
Creatine Kinase myocardial band (U/L) | 0-3 days after randomization (during hospitalization)
  Changes in blood biomarkers
Troponin T in nanogram per millilitre (ng/mL) | 0-3 days after randomization (during hospitalization)
  Changes in blood biomarkers
N-terminal prohormone of brain natriuretic peptide (NT-proBNP) (ng/L) | 0-5 days after randomization (during hospitalization)
  Changes in blood biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Pim van der Harst, Prof. dr., Principal Investigator — University Medical Center Groningen
Locations (3):
- Netherlands (3):
  - Treant Scheper Hospital, Emmen, Drenthe
  - University Medical Centre Groningen, Groningen
  - University Medical Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Koning ML, van Dorp P, Assa S, Hartman MH, Voskuil M, Anthonio RL, Veen D, Pundziute-Do Prado G, Leiner T, van Goor H, van der Meer P, van Veldhuisen DJ, Nijveldt R, Lipsic E, van der Harst P. Rationale and Design of the Groningen Intervention Study for the Preservation of Cardiac Function with Sodium Thiosulfate after St-segment Elevation Myocardial Infarction (GIPS-IV) trial. Am Heart J. 2022 Jan;243:167-176. doi: 10.1016/j.ahj.2021.08.012. Epub 2021 Sep 15. PMID 34534493